CLINICAL TRIAL: NCT06813014
Title: Sitagliptin's Effects on Glucose-stimulated Insulin Secretion and Oral Glucose
Brief Title: Pharmacogenetics of Response to Sitagliptin (PRS)
Acronym: PRS
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Amber Beitelshees, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HP-00111892
Record Dates: First submitted 2025-02-03; First posted 2025-02-06 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Glucose Tolerance Test

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sitagliptin (Experimental): Sitagliptin 100 mg given 2 hours prior to the oral glucose tolerance test
  Interventions: Procedure: Oral Glucose Tolerance Test
- Placebo (Placebo Comparator): Placebo given 2 hours prior to the oral glucose tolerance test
  Interventions: Procedure: Oral Glucose Tolerance Test

INTERVENTIONS:
Procedure: Oral Glucose Tolerance Test — Three hour glucose tolerance test

SUMMARY:
This is a research study to find out how different people respond to a medication called sitagliptin. Sitagliptin is an FDA approved medication that is used to treat diabetes. We are asking for healthy, non-diabetic volunteers to participate in this 7-week study. If you agree to participate, you will take part in 2 clinic visits that are 4-6 weeks apart. At the clinic visits you will have an oral glucose tolerance test (OGTT) and other blood tests to see how your body processes glucose (sugar). An OGTT is a test in which your drink glucose and then blood samples are taken afterward at specific time points to measure glucose and insulin in your blood. Each clinic visit will last about 5 hours.

ELIGIBILITY:
Inclusion Criteria:

* • Age: >18 years old

  * Members of Old Order Amish community in Lancaster, PA

Exclusion Criteria:

* • Pregnancy (reproductive age women will undergo pregnancy tests immediately before receiving the drug)

  * Diabetes: HbA1c > 6.5% or fasting plasma glucose >126 mg/dL
  * Estimated glomerular filtration rates (eGFR) <60 mL/min/1.73 m2
  * Anemia: hematocrit < 35%
  * Thyroid status: TSH<0.4 or TSH>5.5
  * ALT or AST in excess of 2X upper limit of normal
  * Drugs that in the physician's judgment would alter response to sitagliptin
  * Significant health issues that in the physician's judgment could increase the risk for participants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2031-12 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Sitagliptin-induced enhancement of early insulin secretion | 6 weeks
  This represents the incretinomimetic effect of sitagliptin, which contributes importantly to the mechanism whereby DPP4is decrease HbA1c in T2D patients. Because histograms for sitagliptin-induced increase in our index of early insulin secretion (T30:T60) demonstrated a skewed distribution, we will apply a logarithmic transformation of data which yields a normal distribution. Thus, the drug effect is defined as: log(T30:T60 ins)sita - log(T30:T60 ins)control.
Sitagliptin-induced change in glucose tolerance | 6 weeks
  Sitagliptin-induced change in glucose tolerance. This is a consequence of enhanced insulin secretion, which reflects most closely the desired effect of the drug to decrease plasma glucose and decrease HbA1c. Because histograms for sitagliptin-induced increase in our index of glucose tolerance (T30:T60) demonstrated a skewed distribution, we will apply a logarithmic transformation of data which yields a normal distribution. Thus, the drug effect is defined as: log(T30:T60 gluc)sita - log(T30:T60 gluc)control.

SECONDARY OUTCOMES:
Area under the curve for insulin concentration | 6 weeks
  Area under the curve of insulin concentration measured from oral glucose tolerance test using trapezoidal rule
Area under the curve for glucose concentration | 6 weeks
  Area under the curve for glucose concentration measured from the oral glucose tolerance test using the trapezoidal rule
Area under the curve for intact GIP | 6 weeks
  Area under the curve for levels of intact GIP during the first hour of the OGTT as calculated by the trapezoidal rule
Area under the curve for intact GLP1 | 6 weeks
  Area under the curve for levels of intact GLP1 during the first hour of the OGTT as calculated by the trapezoidal rule
Area under the curve for C-peptide levels | 6 weeks
  Area under the curve for C-peptide levels as a direct index of insulin secretion

OTHER OUTCOMES:
Parameters of a mathematical model (insulin secretion and glucose sensitivity of the β-cell | 6 weeks
  We will apply mathematical modeling to the oral glucose tolerance test data it assess measures of insulin secretion and glucose sensitivity of the β-cell

CONTACTS AND LOCATIONS:
Overall Officials: Amber L Beitelshees, PharmD, MPH, Principal Investigator — University of Maryland, Baltimore; Simeon I Taylor, MD, PhD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland Amish Research Clinic, Lancaster, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
Given that the Amish are a unique founder population, they are more easily identified and at-risk for stigmatization. Therefore, we must consult with the community in order to address this plan to share individual level data.